CLINICAL TRIAL: NCT06814041
Title: A Pilot Randomized Controlled Trial and an Interview Study to Evaluate a Chatbot for People Living With HIV in Nigeria
Brief Title: Pilot RCT and Interview Study on an HIV Chatbot in Nigeria
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Pimmer (Other)
Collaborators: University of Ibadan (Other)
Responsible Party: Sponsor-Investigator, Christoph Pimmer, PhD, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IZSTZ0_202602
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: HIV
Keywords: Chatbot; HIV; Nigeria; HIV knowledge; gender
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: The model is: two-arm (1:1), open label, randomised controlled trial (RCT). The intervention group will use the chatbot in addition to the Standard of Care (SoC), the control group will receive SoC only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot Intervention (Experimental): In addition to the Standard of Care described, participants in the intervention group will be able to use a chatbot system. The chatbot was designed especially with the goal to support people newly diagnosed with HIV at the beginning of their antiretroviral therapy (ART).
  Interventions: Other: Chatbot as an informational coach
- Control Group (No Intervention): Study participants in the control group will receive the Standard of Care only, offered by the clinics:
  1. st visit in the clinic: Testing and ART enrolment: When patients in the clinic have a positive HIV test, various health assessments are carried out, including TB testing. The patient has a session with an adherence counsellor. A medical consultation takes place where a doctor addresses health issues and prescribes ART medication. First-time patients receive a 3-month prescription.
  2. nd visit in the clinic in the first three months: Patients return to the clinic within the first 3 months. They are given the results of the tests carried out during their first visit, undergo health checks (vital signs) and receive health information. The patient is also seen by a doctor who prescribes ART for the next 3 months.
  3. rd visit to the clinic at 6 months: The procedure is the same as for the 3-month visit, except that a viral load test is performed.

INTERVENTIONS:
Other: Chatbot as an informational coach — The chatbot acts as an empathic informational coach, performing three main functions: (1) offering short conversation sessions about key topics on living with HIV; (2) responding to users' ad-hoc questions on HIV; (3) reminding users of medical appointments and drug taking.
  The chatbot comprises a conversational system, utilizing WhatsApp for user interaction, with messages routed through the backend Voiceflow. User can access the chatbot system via WhatsApp. That means that they access the chatbot like any other contact in their WhatsApp chat list. The bot incorporates mostly text-based input- and output modalities, and a few images, which are more protective of users' privacy than speech. Concretely, chatbot users interact with the chatbot on WhatsApp by selecting from pre-defined options (buttons) or, in some parts, writing text.
  Arms: Chatbot Intervention

SUMMARY:
This study will investigate the use of a HIV chatbot that acts as an informational coach.

The main question the study aims to answer is:

Does the chatbot improve HIV knowledge in adults (older than 18-years) newly diagnosed with HIV in Nigeria - compared to a control group?

Moreover, the study will also determine potential effects of the chatbot use on patients' resilience, psychological well-being. The study will explore patients' use and perceptions of the chatbot, as well as potential gender differences.

The control group will receive Standard of Care only. Patients in the chatbot intervention group will interact with the chatbot in addition to receiving Standard of Care. They will be able to:

* Use a chatbot via WhatsApp
* Receive information on relevant HIV topics
* Get automated responses to their HIV-related questions
* Be reminded of medical appointments and medication schedules

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HIV
* ART enrollment: at the day of recruitment or in the subsequent 7 days. But no longer than 30 months prior to enrolment in the study..
* Age ≥ 18 years
* Have a personal internet-enabled smartphone with WhatsApp installed
* Carry the phone with them at the time of recruitment
* Able to understand, read, and write in English (the official language in Nigeria)
* Able to understand the information about the study
* Provide written informed consent.

Exclusion Criteria:

* Known pregnancy or ≤3 months postpartum
* Persons with suicidal ideation and/or severe mental distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Participant's HIV knowledge | Baseline to 50-day follow-up
  The primary endpoint is the change of HIV knowledge from baseline to the 50-day follow-up assessed using the Patient's HIV Knowledge Questionnaire (PHKQ). The questionnaire consists of 15 items and includes the components (subscales) Transmission and Misconceptions, Causes and Treatment Outcomes, and Diet and Immunity (Jackson, Okonta, & Ukwe, 2020). Participants are required to evaluate statements such as "HIV infection is caused by evil spirits" using a three-point scale: "Yes," "No," and "I don't know." The correct answer is awarded one point, while incorrect responses or the option "I don't know" are each awarded zero points.

SECONDARY OUTCOMES:
Participants' extended HIV knowledge | at 50 day follow up
  In addition to the Patient's HIV knowledge questionnaire (PHKQ), we will use another knowledge test, which includes 10 additional questions, to more compressively assess the participants' knowledge. The test measures additional knowledge areas, which:
  1. are geared to the study participants' specific situation, i.e. being new to the ART regime (such as how much time it takes until the virus may become undetectable )
  2. are very relevant but not covered by the PHKQ, such as knowing about Post-Exposure-Prophylaxis (PEP) to prevent further infections.
Participants' Resilience (PLHIV Scale) | At 50 day follow up
  To assess whether the availability of an empathic digital agent can also increase people's resilience, i.e. their "positive adaptation within the context of significant adversity", we use the People Living with HIV (PLHIV) Resilience Scale (Gottert et al., 2019). The scale is particularly suited as it is tailored to the situation of people living with HIV, measured and psychometrically validated in three African countries including Uganda, Senegal and Cameroon. The 10-item PLHIV Resilience Scale covers topics such as self-confidence, self-respect etc. and invites participants to indicate whether these have been positively, negatively, or not affected by their HIV status. Higher resilience was associated with less depression in each country (Gottert et al., 2019).
Participants' psychological well-being (SRQ-20) | at 50 day follow up
  Participants' psychological well-being (SRQ-20) - measured at 50 day follow up We will measure participants' psychological well-being with the WHO 20-item Self-Reporting Questionnaire (SRQ-20) (Beusenberg, 1994). SRQ-20 was designed to screen for general psychological distress, especially in developing countries. It contains 20 questions which have to be answered by 'yes' or 'no', such as "are you easily frightened" (Beusenberg, 1994). Scores range from 0 to 20, with higher scores indicating higher levels of distress. SRQ-20 is a widely used and validated measurement to assess psychological distress, including in the context of Nigeria and HIV care. For example, people living with HIV Nigeria were reported to have a thirty-fold increase of psychological distress in the first year on ART (Pierce et al., 2023).
Users' perception of the chatbot: trust and parasocial relationships | at 25 day follow up
  The different ways in which users perceive the chatbot will be measured by assessing users' trust and their perceived relationship with the chatbot.
  Trust is a multidimensional construct and thus a validated measurement tool which consists of three components will be used: competence, benevolence and integrity (Hu & Lu, 2021). Competence consists of 4 items. Benevolence and integrity consist of 3 items each. For example, for benevolence, one question is "whether the digital assistant is interested in my well-being".
  Parasocial relationships questionnaires were originally developed to measure relationships between celebrities and people. They have been applied recently to measure the perceived relational connectedness between chatbots and their users (Youn & Jin, 2021). In this study, the interaction subscale, which consists of 4 items, will be applied. It requires users to evaluate their perceived relationship with the chatbot.

OTHER OUTCOMES:
Chatbot use | 50 day follow up
  Another relevant aspect is to assess usage patterns of the chatbot, especially the intensity of chatbot use. These four main indicators will be extracted from the technical chatbot platform.
  * Number of total interactions per user
  * Number of questions asked per user
  * Number of medication reminders sent to the user
  * Number of conversation topics completed per user
Relationship between sociodemographic characteristics, chatbot use and perception of chatbot, and outcomes: | at 50-day follow up (and for viral load at 6-month follow up)
  The following relationships will be assessed:
  * Relationship between users' gender, age and education status on the one hand side, and chatbot use and chatbot perception at the other hand side
  * Relationship between chatbot use and outcomes (knowledge, resilience, and psychological well-being)
Qualitative goals | about 60 - 90 days after the participant's enrollment, depending on their availability.
  Given the novelty of the intervention in the context at hand, a relevant aspect is to explore the experience of the user to be able to generate an in-depth understanding of the ways in which they perceive the chatbot. This will be achieved through interviews with 15-25 participants from the intervention group. A particular goal of the interviews is to understand whether, and if so, how, female chatbot users perceive the chatbot differently as compared to male users. Trained interviewers will carry out interviews with selected users of the chatbot, i.e. with participants from the intervention group

CONTACTS AND LOCATIONS:
Locations (6):
- Nigeria (6):
  - Infectious Disease Institute, (IDI) UCH, Ibadan, Oyo State
  - St. Mary's Catholic General Hospital, Ibadan, Oyo State
  - Baptist Medical Centre, Saki, Oyo State
  - Adeoyo Maternity Teaching Hospital, Ibadan
  - Our Lady of Apostle Catholic Hospital, Ibadan
  - Ring Road State Hospital, Ibadan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boyd AT, Rocconi LM, Morrow JA. Construct validation and measurement invariance of the Parasocial Relationships in Social Media survey. PLoS One. 2024 Mar 28;19(3):e0300356. doi: 10.1371/journal.pone.0300356. eCollection 2024. PMID 38547192
- [Background] Pierce LJ, Regan S, Idigbe I, Adeola J, Musa Z, Ezechi O, Oladeji B, Gureje O, Freedberg KA, Okonkwo P, Ahonkhai AA. Psychological Distress Increases 30-Fold Among People with HIV in the First Year on ART in Nigeria-a Call for Integrated Mental Health Services. Int J Behav Med. 2023 Feb;30(1):38-48. doi: 10.1007/s12529-022-10068-8. Epub 2022 Feb 28. PMID 35226343
- [Background] Gottert A, Friedland B, Geibel S, Nyblade L, Baral SD, Kentutsi S, Mallouris C, Sprague L, Hows J, Anam F, Amanyeiwe U, Pulerwitz J. The People Living with HIV (PLHIV) Resilience Scale: Development and Validation in Three Countries in the Context of the PLHIV Stigma Index. AIDS Behav. 2019 Sep;23(Suppl 2):172-182. doi: 10.1007/s10461-019-02594-6. PMID 31350712
- [Background] Jackson IL, Okonta JM, Ukwe CV. Development and psychometric evaluation of the patient's HIV knowledge questionnaire (PHKQ). Int J Clin Pharm. 2020 Apr;42(2):695-702. doi: 10.1007/s11096-020-00963-z. Epub 2020 Jan 14. PMID 31939032